CLINICAL TRIAL: NCT05593874
Title: Predictive Value of Nu.Q™ Biomarkers to Help Guiding the Management of Osteoarticular Infections - a Monocentric Prospective Observational Cohort Study
Brief Title: Predictive Value of Nu.Q™ Biomarkers to Help Guiding the Management of Osteoarticular Infections
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Mikael de Lorenzi-Tognon, Principal Subinvestigator, University Hospital, Geneva
Other Study IDs: 2022-00140
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot; Chronic Osteomyelitis; Septic Arthritis
Keywords: diabetic foot; osteoarticular infections
MeSH Terms: conditions — Diabetic Foot; Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Centrifugated blood samples (serum/plasma used for analyses)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic foot ulcer with osteoarticular infections: Diabetic patients suffering from ulcer that led to an osteoarticular infection (e.g. chronic osteomyelitis, septic arthritis)
  Interventions: Diagnostic Test: Histones H3.1 blood levels

INTERVENTIONS:
Diagnostic Test: Histones H3.1 blood levels — Measure of blood concentrations of histone subtype H3.1

SUMMARY:
Diabetic foot ulcers are frequent with average lifetime risk of 15%, and can lead to bone and joint infections. Current protocols for their management include evaluation of ischemia, assessment of underlying bone infection, sharp debridement, off-loading and use of dressings that promote moist wound healing. Extensive debridement is optimal for wound healing and decreases the risk of recurrence. However, extension of surgical debridement is left at the clinician judgement and thus lacks standardised protocols. Plus, there is currently no known risk factors or specific biomarkers that can help guide the clinician for the extent of debridement or that can predict a recurrence in case of non-extensive debridement. The main objectives of the study are to either unravel a new biomarker, and/or identify risk factors associated with poor prognosis following surgical debridement in diabetic foot ulcers. Histones, more specifically H3.1 subtype, have been associated with sepsis.

The main hypothesis is that higher blood levels of H3.1 will be present in participants showing poor prognosis (i.e., having additional surgeries, amputation, death) and that a rise in H3.1 blood levels compared to baseline (before the 1st surgical intervention) would provide an early warning of relapse or treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years old) suffering from diabetes mellitus (type 1 or 2)
* Diabetic foot ulcer with severe infection (grade 3 and 4 according to IWGDF 2019 classification)
* Scheduled surgical debridement

Exclusion Criteria:

* Spondylodiscitis
* Pregnant or lactating women
* Previous enrolment in a clinical trial
* Consent declined by participant or tutor in case of incapacitation
* Tutor cannot be reached for consent in case of incapacitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All diabetic patients fulfilling the inclusion criteria with no exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Clinical failure | day 30 and day 60
  Presence of infection (IWGDF 2019 criteria) and No change in H3.1 blood levels from baseline (day -1) or secondary increase after an initial decline ≥ 75%

SECONDARY OUTCOMES:
Mortality | day 30 and day 60
  Death during the study period from day-1 (day of the 1st intervention)
Amputation rate | day 1 to day 60
  Frequency of the event 'amputation' as incidence rate from day-1 (day of the 1st intervention)
Additional surgical interventions rate | day 1 to day 60
  Frequency of the event 'additional surgical intervention' (i.e., debridement, amputation) as incidence rate from day-1 (day of the 1st intervention)
Time-to-amputation | day 1 to day 60
  Measured in days from day-1 (day of the 1st intervention)
Time-to-additional-intervention | day 1 to day 60
  Measured in days from day-1 (day of the 1st intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monteiro-Soares M, Russell D, Boyko EJ, Jeffcoate W, Mills JL, Morbach S, Game F; International Working Group on the Diabetic Foot (IWGDF). Guidelines on the classification of diabetic foot ulcers (IWGDF 2019). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3273. doi: 10.1002/dmrr.3273. PMID 32176445
- [Background] Lebrun E, Tomic-Canic M, Kirsner RS. The role of surgical debridement in healing of diabetic foot ulcers. Wound Repair Regen. 2010 Sep-Oct;18(5):433-8. doi: 10.1111/j.1524-475X.2010.00619.x. PMID 20840517
- [Background] Thiam HR, Wong SL, Qiu R, Kittisopikul M, Vahabikashi A, Goldman AE, Goldman RD, Wagner DD, Waterman CM. NETosis proceeds by cytoskeleton and endomembrane disassembly and PAD4-mediated chromatin decondensation and nuclear envelope rupture. Proc Natl Acad Sci U S A. 2020 Mar 31;117(13):7326-7337. doi: 10.1073/pnas.1909546117. Epub 2020 Mar 13. PMID 32170015
- [Background] Wong SL, Demers M, Martinod K, Gallant M, Wang Y, Goldfine AB, Kahn CR, Wagner DD. Diabetes primes neutrophils to undergo NETosis, which impairs wound healing. Nat Med. 2015 Jul;21(7):815-9. doi: 10.1038/nm.3887. Epub 2015 Jun 15. PMID 26076037
- [Background] Li Y, Liu B, Fukudome EY, Lu J, Chong W, Jin G, Liu Z, Velmahos GC, Demoya M, King DR, Alam HB. Identification of citrullinated histone H3 as a potential serum protein biomarker in a lethal model of lipopolysaccharide-induced shock. Surgery. 2011 Sep;150(3):442-51. doi: 10.1016/j.surg.2011.07.003. PMID 21878229
- [Background] Eichhorn T, Linsberger I, Laukova L, Tripisciano C, Fendl B, Weiss R, Konig F, Valicek G, Miestinger G, Hormann C, Weber V. Analysis of Inflammatory Mediator Profiles in Sepsis Patients Reveals That Extracellular Histones Are Strongly Elevated in Nonsurvivors. Mediators Inflamm. 2021 Mar 17;2021:8395048. doi: 10.1155/2021/8395048. eCollection 2021. PMID 33790693
- [Background] Morimont L, Dechamps M, David C, Bouvy C, Gillot C, Haguet H, Favresse J, Ronvaux L, Candiracci J, Herzog M, Laterre PF, De Poortere J, Horman S, Beauloye C, Douxfils J. NETosis and Nucleosome Biomarkers in Septic Shock and Critical COVID-19 Patients: An Observational Study. Biomolecules. 2022 Jul 27;12(8):1038. doi: 10.3390/biom12081038. PMID 36008932